CLINICAL TRIAL: NCT04318587
Title: Assessment of Donor Derived Cell Free DNA and Utility in Lung Transplantation
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Due to COVID and staffing shortages we decided to end the study with 40 participants instead of 50.
Sponsor: Pablo Sanchez (Other)
Collaborators: CareDx (Industry)
Responsible Party: Sponsor-Investigator, Pablo Sanchez, Vice Chair, Benign Lung Diseases Surgical Director, Lung Transplant and ECMO, Director, Lung Transplant Research and ELVP Program, University of Pittsburgh
Organization: University of Pittsburgh (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: STUDY19090098
Record Dates: First submitted 2020-03-17; First posted 2020-03-24 (Actual); Results first posted 2024-03-25 (Actual); Last update posted 2024-03-25 (Actual); Status verified 2024-03

CONDITIONS: Lung Transplant Failure and Rejection
MeSH Terms: conditions — Rejection, Psychology

STUDY DESIGN:
Intervention Model Description: Correlate donor DNA in blood samples to episodes of Acute rejection diagnosed by transbronchial biopsy and BOS/CLAD diagnosed by spirometry
  From this correlation we hope to be able to develop a miniMally invasive test ( blood sample) that can predict or correlate acute and or chronic rejection
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (1):
- Allosure Arm (Experimental): All subjects will be in arm one and will have AlloSure blood draws at multiple time points.
  Interventions: Diagnostic Test: Allosure

INTERVENTIONS:
Diagnostic Test: Allosure — Blood is collected from the patient, packaged, and shipped at ambient temperature to CareDx for testing. Donor-derived cell-free DNA is measured via targeted amplification and sequencing of a set of carefully selected and validated SNPs. The AlloSure bioinformatics software calculates the percent dd-cfDNA in the sample tested and applies the QC criteria. The AlloSure results will be compared to the episodes of acute rejection diagnosed by transbronchial biopsy and BOS/CLAD diagnosed by spirometry in the subjects medical records. Transbronchial biopsies and spirometry are standard of care for lung transplant recipients.

SUMMARY:
The use of Allosure to identify and quantify circulating donor-derived cell-free DNA to quantitate allograft injury in the early post-transplant period and determine its relationship to allograft failure.

DETAILED DESCRIPTION:
Single Center Prospective Cohort Study on De-Novo Lung Transplant recipients. AlloSure will be drawn as part of routine blood draws and sent to CareDx for analysis of dd-cfDNA. All data will be collected and stored in the hospital EMR, this will be examined with the AlloSure results to correlate outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Participant is willing and able to give informed consent for participation in the study.
* Male or Female, aged 18 years or above.
* Denovo lung transplant recipient
* Ability to understand written and spoken English

Exclusion Criteria:

* Previous transplant or multi-organ transplant
* Unable to have blood draw for medical reason

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2020-06-29 (Actual); Primary Completion 2022-12-31 (Actual); Study Completion 2023-12-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pablo Sanchez, MD, Principal Investigator — Associate Program Director Residency Program
Locations (1):
- UPMC Presbyterian, Pittsburgh, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data that underlie the results reported in the article, after de-identification (text, tables, figures, and appendices)
Supporting Information: Study Protocol
Time Frame: Beginning 9 months and ending 36 months following article publication
Access Criteria: Investigators whose proposed use of the data has been approved by an independent review committee identified for this purpose.

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Allosure Arm
Started | 40
Completed | 40
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Allosure Arm
Number analyzed (Participants) | 40
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 26
  >=65 years | 14
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 17
  Male | 23
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 40

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Primary Graft Dysfunction/Allograft Rejection 24 Hours Post Transplant
Description: Primary Graft Dysfunction is measured using a combination of radiographic opacification and P:F ratio (ratio of partial pressure of oxygen related to fraction of inhaled oxygen).
  Grade 0: No opacifications on CXR Grade 1: Opacifications and P:F > 300 Grade 2: Opacifications and P:F >200, < 300 Grade 3: Opacifications and P:F < 200
  If someone requires ECMO, they are automatically a grade 3.
Time Frame: 24 hours post transplant
Measure: Count of Participants; unit: Participants
Arm/Group | Allosure Arm
Number analyzed (Participants) | 40
Participants
  PGD 1 | 15
  PGD 2 | 2
  PGD 3 | 8

2. Primary Outcome: Number of Participants With Primary Graft Dysfunction/Allograft Rejection 48 Hours Post Transplant
Description: as for outcome 1
Time Frame: 48 hours post transplant
Measure: Count of Participants; unit: Participants
Arm/Group | Allosure Arm
Number analyzed (Participants) | 40
Participants
  PGD 1 | 19
  PGD 2 | 1
  PGD 3 | 10

3. Primary Outcome: Number of Participants With Primary Graft Dysfunction/Allograft Rejection 72 Hours Post Transplant
Description: as for outcome 1
Time Frame: 72 hours post transplant
Measure: Count of Participants; unit: Participants
Arm/Group | Allosure Arm
Number analyzed (Participants) | 40
Participants
  PGD 1 | 15
  PGD 2 | 1
  PGD 3 | 11

4. Primary Outcome: Number of Participants With Allograft Rejection 3 Months Post Transplant
Description: Number of participants that experienced allograft rejection determined by evaluation of biopsy taken during bronchoscopy.
Time Frame: 3 months post transplant
Measure: Count of Participants; unit: Participants
Arm/Group | Allosure Arm
Number analyzed (Participants) | 40
Participants | 6

5. Primary Outcome: Number of Participants With Allograft Rejection 6 Months Post Transplant
Description: as for outcome 4
Time Frame: 6 months post transplant
Measure: Count of Participants; unit: Participants
Arm/Group | Allosure Arm
Number analyzed (Participants) | 40
Participants | 0

6. Primary Outcome: Number of Participants With Allograft Rejection 9 Months Post Transplant
Description: as for outcome 4
Time Frame: 9 months post transplant
Measure: Count of Participants; unit: Participants
Arm/Group | Allosure Arm
Number analyzed (Participants) | 40
Participants | 0

7. Primary Outcome: Number of Participants With Allograft Rejection 12 Months Post Transplant
Description: as for outcome 4
Time Frame: 12 months post transplant
Measure: Count of Participants; unit: Participants
Arm/Group | Allosure Arm
Number analyzed (Participants) | 40
Participants | 0

8. Primary Outcome: Amount of Allosure Donor Derived Cell Free DNA (Dd-cDNA) Pre-Transplant
Description: dd-cDNA is fragmented DNA that originates from cells and is released into the bloodstream. This fragmented DNA is donor/recipient specific. The Allosure test is able to measure the specific amount of DNA derived from the donor cells.
  Amount of Allosure Donor Derived Cell Free DNA (dd-cDNA) Pre-Transplant
Time Frame: pre-transplant
Measure: Mean (Standard Deviation); unit: %dd-cfDNA
Arm/Group | Allosure Arm
Number analyzed (Participants) | 34
%dd-cfDNA | 0.014 (0.05)

9. Primary Outcome: Amount of Allosure Donor Derived Cell Free DNA (Dd-cDNA) 24 Hours Post Transplant
Description: dd-cDNA is fragmented DNA that originates from cells and is released into the bloodstream. This fragmented DNA is donor/recipient specific. The Allosure test is able to measure the specific amount of DNA derived from the donor cells.
Time Frame: 24 hours post-transplant
Measure: Mean (Standard Deviation); unit: %dd-cfDNA
Arm/Group | Allosure Arm
Number analyzed (Participants) | 34
%dd-cfDNA | 15.4 (4.5)

10. Primary Outcome: Amount of Allosure Donor Derived Cell Free DNA (Dd-cDNA) 48 Hours Post Transplant
Description: as for outcome 9
Time Frame: 48 hours post-transplant
Measure: Mean (Standard Deviation); unit: %dd-cfDNA
Arm/Group | Allosure Arm
Number analyzed (Participants) | 35
%dd-cfDNA | 11.56 (5.23)

11. Primary Outcome: Amount of Allosure Donor Derived Cell Free DNA (Dd-cDNA) 72 Hours Post Transplant
Description: as for outcome 9
Time Frame: 72 hours post-transplant
Measure: Mean (Standard Deviation); unit: %dd-cfDNA
Arm/Group | Allosure Arm
Number analyzed (Participants) | 35
%dd-cfDNA | 8.41 (3.85)

12. Primary Outcome: Amount of Allosure Donor Derived Cell Free DNA (Dd-cDNA) 1 Week Post Transplant
Description: as for outcome 9
Time Frame: 1 week post-transplant
Measure: Mean (Standard Deviation); unit: %dd-cfDNA
Arm/Group | Allosure Arm
Number analyzed (Participants) | 37
%dd-cfDNA | 5.08 (2.30)

13. Primary Outcome: Amount of Allosure Donor Derived Cell Free DNA (Dd-cDNA) 2 Weeks Post Transplant
Description: dd-cDNA is fragmented DNA that originates from cells and is released into the bloodstream. This fragmented DNA is donor/recipient specific. The Allosure test is able to measure the specific amount of DNA derived from the donor cells.
  Amount of Allosure Donor Derived Cell Free DNA (dd-cDNA) 2 Weeks Post Transplant
Time Frame: 2 weeks post-transplant
Measure: Mean (Standard Deviation); unit: %dd-cfDNA
Arm/Group | Allosure Arm
Number analyzed (Participants) | 35
%dd-cfDNA | 4.84 (16.04)

14. Primary Outcome: Amount of Allosure Donor Derived Cell Free DNA (Dd-cDNA) 3 Weeks Post Transplant
Description: as for outcome 9
Time Frame: 3 weeks post-transplant
Measure: Mean (Standard Deviation); unit: %dd-cfDNA
Arm/Group | Allosure Arm
Number analyzed (Participants) | 29
%dd-cfDNA | 2.32 (1.35)

15. Primary Outcome: Amount of Allosure Donor Derived Cell Free DNA (Dd-cDNA) 4 Weeks Post Transplant
Description: as for outcome 9
Time Frame: 4 weeks post-transplant
Measure: Mean (Standard Deviation); unit: %dd-cfDNA
Arm/Group | Allosure Arm
Number analyzed (Participants) | 20
%dd-cfDNA | 2.58 (2.09)

16. Primary Outcome: Amount of Allosure Donor Derived Cell Free DNA (Dd-cDNA) 5 Weeks Post Transplant
Description: as for outcome 9
Time Frame: 5 weeks post-transplant
Measure: Mean (Standard Error); unit: %dd-cfDNA
Arm/Group | Allosure Arm
Number analyzed (Participants) | 23
%dd-cfDNA | 2.09 (1.33)

17. Primary Outcome: Amount of Allosure Donor Derived Cell Free DNA (Dd-cDNA) 6 Weeks Post Transplant
Description: as for outcome 9
Time Frame: 6 weeks post-transplant
Measure: Mean (Standard Deviation); unit: %dd-cfDNA
Arm/Group | Allosure Arm
Number analyzed (Participants) | 15
%dd-cfDNA | 1.43 (0.87)

18. Primary Outcome: Amount of Allosure Donor Derived Cell Free DNA (Dd-cDNA) 7 Weeks Post Transplant
Description: as for outcome 9
Time Frame: 7 weeks post-transplant
Measure: Mean (Standard Deviation); unit: %dd-cfDNA
Arm/Group | Allosure Arm
Number analyzed (Participants) | 14
%dd-cfDNA | 1.06 (0.67)

19. Primary Outcome: Amount of Allosure Donor Derived Cell Free DNA (Dd-cDNA) 8 Weeks Post Transplant
Description: as for outcome 9
Time Frame: 8 weeks post-transplant
Measure: Mean (Standard Deviation); unit: %dd-cfDNA
Arm/Group | Allosure Arm
Number analyzed (Participants) | 9
%dd-cfDNA | 0.91 (0.49)

20. Primary Outcome: Amount of Allosure Donor Derived Cell Free DNA (Dd-cDNA) 9 Weeks Post Transplant
Description: as for outcome 9
Time Frame: 9 weeks post-transplant
Measure: Mean (Standard Deviation); unit: %dd-cfDNA
Arm/Group | Allosure Arm
Number analyzed (Participants) | 14
%dd-cfDNA | 0.85 (0.50)

21. Primary Outcome: Amount of Allosure Donor Derived Cell Free DNA (Dd-cDNA) 10 Weeks Post Transplant
Description: as for outcome 9
Time Frame: 10 weeks post-transplant
Measure: Mean (Standard Deviation); unit: %dd-cfDNA
Arm/Group | Allosure Arm
Number analyzed (Participants) | 14
%dd-cfDNA | 0.74 (0.49)

22. Primary Outcome: Amount of Allosure Donor Derived Cell Free DNA (Dd-cDNA) 11 Weeks Post Transplant
Description: as for outcome 9
Time Frame: 11 weeks post-transplant
Measure: Mean (Standard Deviation); unit: %dd-cfDNA
Arm/Group | Allosure Arm
Number analyzed (Participants) | 11
%dd-cfDNA | 0.89 (0.49)

23. Primary Outcome: Amount of Allosure Donor Derived Cell Free DNA (Dd-cDNA) 12 Weeks Post Transplant
Description: as for outcome 9
Time Frame: 12 weeks post-transplant
Measure: Mean (Standard Deviation); unit: %dd-cfDNA
Arm/Group | Allosure Arm
Number analyzed (Participants) | 14
%dd-cfDNA | 1.04 (1.01)

24. Primary Outcome: Amount of Allosure Donor Derived Cell Free DNA (Dd-cDNA) 4 Months Post Transplant
Description: as for outcome 9
Time Frame: 4 months post transplant
Measure: Mean (Standard Deviation); unit: %dd-cfDNA
Arm/Group | Allosure Arm
Number analyzed (Participants) | 16
%dd-cfDNA | 0.85 (1.04)

25. Primary Outcome: Amount of Allosure Donor Derived Cell Free DNA (Dd-cDNA) 5 Months Post Transplant
Description: as for outcome 9
Time Frame: 5 months post transplant
Measure: Mean (Standard Deviation); unit: %dd-cfDNA
Arm/Group | Allosure Arm
Number analyzed (Participants) | 15
%dd-cfDNA | 0.67 (0.53)

26. Primary Outcome: Amount of Allosure Donor Derived Cell Free DNA (Dd-cDNA) 6 Months Post Transplant
Description: as for outcome 9
Time Frame: 6 months post-transplant
Measure: Mean (Standard Deviation); unit: %dd-cfDNA
Arm/Group | Allosure Arm
Number analyzed (Participants) | 16
%dd-cfDNA | 0.92 (0.86)

27. Primary Outcome: Amount of Allosure Donor Derived Cell Free DNA (Dd-cDNA) 7 Months Post Transplant
Description: as for outcome 9
Time Frame: 7 months post-transplant
Measure: Mean (Standard Deviation); unit: %dd-cfDNA
Arm/Group | Allosure Arm
Number analyzed (Participants) | 8
%dd-cfDNA | 1.01 (1.58)

28. Primary Outcome: Amount of Allosure Donor Derived Cell Free DNA (Dd-cDNA) 8 Months Post Transplant
Description: as for outcome 9
Time Frame: 8 months post-transplant
Measure: Mean (Standard Deviation); unit: %dd-cfDNA
Arm/Group | Allosure Arm
Number analyzed (Participants) | 8
%dd-cfDNA | 0.50 (0.58)

29. Primary Outcome: Amount of Allosure Donor Derived Cell Free DNA (Dd-cDNA) 9 Months Post Transplant
Description: as for outcome 9
Time Frame: 9 months post-transplant
Measure: Mean (Standard Deviation); unit: %dd-cfDNA
Arm/Group | Allosure Arm
Number analyzed (Participants) | 5
%dd-cfDNA | 0.92 (0.66)

30. Primary Outcome: Amount of Allosure Donor Derived Cell Free DNA (Dd-cDNA) 10 Months Post Transplant
Description: as for outcome 9
Time Frame: 10 months post-transplant
Measure: Mean (Standard Deviation); unit: %dd-cfDNA
Arm/Group | Allosure Arm
Number analyzed (Participants) | 7
%dd-cfDNA | 0.67 (0.61)

31. Primary Outcome: Amount of Allosure Donor Derived Cell Free DNA (Dd-cDNA) 11 Months Post Transplant
Description: as for outcome 9
Time Frame: 11 months post-transplant
Measure: Mean (Standard Deviation); unit: %dd-cfDNA
Arm/Group | Allosure Arm
Number analyzed (Participants) | 8
%dd-cfDNA | 0.67 (0.39)

32. Primary Outcome: Amount of Allosure Donor Derived Cell Free DNA (Dd-cDNA) 12 Months Post Transplant
Description: as for outcome 9
Time Frame: 12 months post-transplant
Measure: Mean (Standard Deviation); unit: %dd-cfDNA
Arm/Group | Allosure Arm
Number analyzed (Participants) | 16
%dd-cfDNA | 0.56 (0.83)

33. Secondary Outcome: Number of Participants That Experienced Graft Failure or Death Within One Year Post Transplant
Description: The number of participants that were diagnosed as having chronic lung allograft dysfunction (CLAD), needed re-transplanted or died before 1 year post transplant.
Time Frame: one year post transplant
Measure: Count of Participants; unit: Participants
Arm/Group | Allosure Arm
Number analyzed (Participants) | 40
Participants | 0

ADVERSE EVENTS:
Time Frame: 1 year
Arm/Group | Allosure Arm
All-Cause Mortality (participants affected / at risk) | 3/40
Serious Adverse Events (participants affected / at risk) | 0/40
Other Adverse Events (participants affected / at risk) | 0/40

LIMITATIONS AND CAVEATS:
Not every patient had blood collected at the specified time points. Blood was missed at time of bronchoscopy or patient cancelled their bronchoscopy. 515 blood samples drawn and shipped to CareDx. 2 samples lost after they arrived at CareDx. Of the 513 samples assessed, we were not able to get the %dd-cfDNA data for 36 samples. This was due to sample quality and assay quality metrics. Hemolysis was the main reason for incomplete data.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-06-27): https://cdn.clinicaltrials.gov/large-docs/87/NCT04318587/Prot_SAP_000.pdf